CLINICAL TRIAL: NCT06382467
Title: Comparison of Remimazolam and Propofol Combination vs. Propofol in Intraoperative Neurophysiologic Monitoring: A Randomized Controlled Trial
Brief Title: Comparison of Remimazolam and Propofol Combination vs. Propofol in IOM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Gwangmyeong Hospital (Other)
Responsible Party: Principal Investigator, Jiwon Han, Assistant professor, Chung-Ang University Gwangmyeong Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2401-136-016
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination group (Experimental): Combination regimen (remimazolam plus propofol)
  Interventions: Drug: Remimazolam besylate + propofol MCT
- Propofol group (Active Comparator): Propofol monotherapy
  Interventions: Drug: Propofol MCT

INTERVENTIONS:
Drug: Remimazolam besylate + propofol MCT — remimazolam besylate 3mg/kg/hr for induction, and 0.5 mg/kg/hr for maintenance + propofol MCT 1-4 mcg/ml using target-controlled infusion
  Arms: Combination group
Drug: Propofol MCT — Propofol MCT 2-8 mcg/ml using target-controlled infusion
  Arms: Propofol group

SUMMARY:
This study aims to compare total intravenous anesthetic agents: combined remimazolam and propofol vs. propofol monotherapy. The comparison parameters are intraoperative hypotension, patient's involuntary movement, neurophysiological monitoring quality, onset time, recovery time, and postoperative rescue anti-emetics requirements.

DETAILED DESCRIPTION:
This study hypothesizes that the combination regimen of remimazolam and propofol as total intravenous anesthesia in neurosurgical procedures requiring neurophysiological monitoring can reduce the incidence of hypotension compared to propofol monotherapy while providing comparable levels of neurophysiological monitoring and surgical conditions. With this hypothesis, the study aims to compare the frequency, severity, and duration of hypotension, frequency of patient movement, and appropriateness of neurophysiological monitoring between the combination therapy of remimazolam and propofol and propofol monotherapy in total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 and above with planned neurosurgical procedures requiring neurophysiological monitoring, classified as American Society of Anesthesiologists (ASA) physical status classification 1, 2, or 3 in the United States.

Exclusion Criteria:

1. Patients who refuse to participate in the study.
2. Patients who are pregnant or lactating.
3. Patients with hypersensitivity to the investigational drugs or to soy, peanuts, or Dextran 40.
4. Patients with acute narrow-angle glaucoma.
5. Patients with alcohol or drug dependence.
6. Patients with hepatic impairment classified as Child-Pugh class C.
7. Patients with lactose intolerance.
8. Patients requiring emergency surgery.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | operation day - postoperative 1 day
  mean arterial pressure < 65mmHg

SECONDARY OUTCOMES:
Amount and number of inotropic agents | operation day - postoperative 1 day
  intraoperative inotropics amount (phenylephrine(mcg), ephedrine(mg), norepinephrine(mcg), dopamine(mg))
Incidence of participants' intraoperative involuntary movement | operation day - postoperative 1 day
  number of patients involuntary movement during operation (ex. no movement:0 , 3 times of movement: 3)
scores of neurophysiologic monitoring quality | operation day - postoperative 1 day
  0-5 scale of neurophysiologic monitoring quality, scored by neurophysiologic monitoring technologist (poor: 0, good: 5)
onset time of study drugs | operation day - postoperative 1 day
  time from administration of study drugs(remimazolam+propofol or propofol) to Bispectral index value < 60
The administration number of rescue anti-emetic agents | operation day - postoperative 3 day
  postoperative rescue anti-emetic agents (ramosetron, palonosetron, metoclopramide) requirements
Time-weighted average of intraoperative hypotension | operation day - postoperative 1 day
  (depth of hypotension in millimeters of mercury below a MAP of 65mmHg × time in minutes spent below a MAP of 65mmHg)÷total duration of operation in minutes
recovery time of study drugs (remimazolam+propofol or propofol) | operation day - postoperative 1 day
  time from discontinuation of study drugs(remimazolam+propofol or propofol) to Bispectral index value > 60

IPD SHARING:
Plan to Share IPD: Undecided